CLINICAL TRIAL: NCT05244343
Title: Impact of Vaccination on Medical and Intensive Care Hospitalization of COVID-19 Patients
Brief Title: I VACCIN Hospitalization of COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Eshmoun Clinical Research Center (Network)
Responsible Party: Sponsor
Other Study IDs: I VACCIN
Record Dates: First submitted 2022-02-16; First posted 2022-02-17 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: SARS CoV 2 Infection; COVID-19
Keywords: COVID-19; Vaccination; Hospitalization
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A REALLIFE evaluation of rate of hospitalized patients in Intensive Care Units and in medical Units of non -vaccinated patients vs vaccinated patients

DETAILED DESCRIPTION:
Transversal National multicenter non interventional on the COVID-19 vaccines

* Period of hospitalization: from January 1st to March 3rd, 2022
* Recruitment duration: 37 days
* Total study duration: 44 days

ELIGIBILITY:
Inclusion Criteria:

* Male and Female ≥ 18 years
* Confirmed COVID-19 patients hospitalized in ICU and Medical Units during the period of the study from January 1st to March 3rd.

Exclusion Criteria:

* Subjects vaccinated outside Tunisia
* Subjects <18 years
* Not confirmed COVID-19
* Not hospitalized patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized due to COVID-19 in ICU or medical units, who are ≥ 18 years old during the period extended from January 1st to March 3rd.
Sampling Method: Non-Probability Sample
Enrollment: 1096 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Rate of COVID-19 not vaccinated patients hospitalized in ICU | From January 1st to February 15th
  Rate of non vaccinated patients who were hospitalized in ICU due to COVID-19 compared to all patients hospitalized due to COVID-19
Rate of COVID-19 not fully vaccinated patients hospitalized in ICU | From January 1st to February 15th
  Rate of not fully vaccinated patients who were hospitalized in ICU due to COVID-19 compared to the total number of Hospitalized patients

SECONDARY OUTCOMES:
Rate of COVID-19 not vaccinated patients hospitalized in Medical Units | From January 1st to February 15th
  Rate of non vaccinated patients who were hospitalized in Medical units due to COVID-19 compared to all patients hospitalized due to COVID-19
Rate of COVID-19 not fully vaccinated patients hospitalized in Medical Units | From January 1st to February 15th
  Rate of not fully vaccinated patients who were hospitalized in Medical units due to COVID-19 compared to all patients hospitalized due to COVID-19
Rate of COVID-19 vaccinated patients hospitalized in Medical Unit by type of vaccine | From January 1st to February 15th
  Rate of COVID-19 vaccinated patients hospitalized in Medical Unit by type of vaccine received

CONTACTS AND LOCATIONS:
Overall Officials: Mariem Melliti, Study Director — Eshmoun Clinical Research Center
Locations (1):
- Abderrahmen Mami Hospital, Aryanah, Tunisia

IPD SHARING:
Plan to Share IPD: No